CLINICAL TRIAL: NCT05209048
Title: Risk Factors and a Nomogram of Venous Thromboembolism in Adult Patients After Orthotopic Liver Transplantation Base on a Single-center Case-control Study
Brief Title: Risk Factors and a nOmogram of Venous thromboEmbolism in Patients After liveR Transplantation(ROVER Study)
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 19242-401
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-12

CONDITIONS: Venous Thromboembolism; Liver Transplantation
Keywords: VTE; OLT; Risk factor; Nomogram model
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- VTE of Derivation group: VTE of Derivation group includes patients who underwent orthotopic liver transplantation on 2018.8-2020.12 and developed VTE within 30 days after operation
- No-VTE of Derivation group: No-VTE of Derivation group includes patients who underwent orthotopic liver transplantation on 2018.8-2020.12 and did not develop VTE within 30 days after surgery or after 30 days
- VTE of Validation group: VTE of Validation group includes patients who underwent orthotopic liver transplantation on 2021.1-2021.12 and developed VTE within 30 days after operation
- No-VTE of Validation group: No-VTE of Validation group includes patients who underwent orthotopic liver transplantation on 2021.1-2021.12 and did not develop VTE within 30 days after surgery or after 30 days

SUMMARY:
Liver transplantation is currently an effective treatment for end-stage liver disease. The high incidence of thrombotic related complications in the early postoperative period after orthotopic liver transplantation(OLT) has been attributed to many factors, such as the long operation time, the high trauma, the need for prolonged bed rest after operation, and the instability of coagulation status in the early postoperative period. Among them, venous thromboembolism (VTE) is one of the most common complications after liver transplantation, including deep vein thrombosis (DVT) and pulmonary embolism (PE), which seriously affect the survival of patients after transplantation. Although the Caprini score is currently recognized as a more mature thrombotic risk assessment tool in patients undergoing abdominal surgery. However, because of the long operation time of liver transplantation and central venous catheterization and other factors, the majority of surgical patients score ≥ 5 points, which are all very high-risk grades. It loses the power of this model for risk stratification and targeted prevention. How to correctly identify people at high risk of VTE after OLT, early diagnosis of VTE and aggressive implementation of correct preventive measures appear essential. Therefore, this study was designed as a single center case-control study to review and analyze the incidence, clinical characteristics, and associated risk factors of VTE after OLT, and to establish a nomogram risk assessment model and validate its predictive efficacy.

DETAILED DESCRIPTION:
In this study, the investigators recruited adult inpatients who underwent orthotopic liver transplantation at Tsinghua Chang Gung Memorial Hospital, Beijing, from August 2018 to December 2021. The hospitalized patients who developed VTE within 30 days after liver transplantation were screened according to the inclusion and exclusion criteria, and similarly, the negative patients were those who did not develop VTE perioperatively or who developed VTE greater than 30 days postoperatively. The diagnosis of VTE was confirmed as the occurrence of a critical value alert during hospitalization, which was predefined as ultrasound/radiology report of DVT or/and PE. Data were obtained from the medical record bank of Tsinghua Chang Gung Memorial Hospital, affiliated to Tsinghua University, Beijing, China. Patient general data, laboratory test data, surgical information, etc. were extracted from the database. To analyze the incidence, clinical characteristics, and risk factors of VTE in patients after liver transplantation. Based on risk factors, a risk assessment model was built with liver transplant inpatient data from August 2018 to December 2020, and the model was validated with liver transplant inpatient data from January 2021 to December 2021.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. With orthotopic whole-liver transplantation
3. Liver was obtained from Brain-dead organ donors

Exclusion Criteria:

1. Living donor liver transplantation, split liver transplantation, partial donor liver transplantation
2. Multivisceral or combined organ transplantation
3. Patients with preoperative VTE
4. Age < 18 years
5. Died or discontinued surgery during surgery
6. Those who died within 48 h after surgery or were discharged from hospital on their own resulting treatment discontinuity
7. Patients with incomplete clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators recruited adult inpatients who received whole liver orthotopic liver transplantation in Beijing Tsinghua Changgeng hospital from August 2018 to December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The rate of VTE after OLT | From August 2018 to December 2021
  The diagnosis of VTE was confirmed as the occurrence of a critical value alert during hospitalization, which was predefined as ultrasound/radiology report of DVT or/and PE.

SECONDARY OUTCOMES:
Patients' preoperative general information | From August 2018 to December 2021
  The general preoperative information of the patients included gender, age, etiology, BMI, comorbidities (hypertension, diabetes mellitus, coronary heart disease, hyperlipidemia, and history of renal insufficiency), surgical history, etc
Perioperative laboratory test indicators of patients | From August 2018 to December 2021
  Laboratory test data: total bilirubin (TBIL), direct bilirubin (DBIL), alanine aminotransferase (ALT), glutamic oxalacetic transaminase (AST) glutamyltransferase (GGT), serum creatinine (SCR), serum albumin (ALB), platelet count (PLT), hemoglobin (HB), D-Dimer (D-dimer), international normalized ratio (INR), prothrombin time (APTT), etc. D-dimer was serially collected from preoperatively to 2 weeks postoperatively. For the remaining items, the test data were collected preoperatively, on postoperative day 1, and on postoperative day 7
Surgical information | From August 2018 to December 2021
  Surgical information included operative method, intraoperative blood loss, plasma transfusion, red blood cell transfusion, prothrombin complex amount, liver free period time, low central venous pressure (CVP ≤ 5 cm H2O) time, operative time, ASA score, model for end stage liver disease (MELD) score, postoperative ICU stay, caprini score

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Wu, MD, Principal Investigator — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hosipital, Beijing, Beijing Municipality, China